CLINICAL TRIAL: NCT01186978
Title: Dose-Reduced Consolidation Radiation Therapy in Patients With Diffuse Large B-cell Lymphoma
Brief Title: Reduced Radiation in Patients With Diffuse Large B-cell Lymphoma
Acronym: DLBCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025164
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): This phase II study will evaluate whether a reduction in the RT dose, concomitant with a decrease in the RT field size, in patients that achieve CR and have a negative post-chemotherapy PET scan following 4 to 6 cycles of rituximab containing chemotherapy, will be associated with a low risk of in-field failure. The goal of this approach is to maintain excellent control rates while minimizing the risk of acute and late toxicity.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — 1.5-2 Gy per fraction to a total dose of 19.8-20 Gy with radiation given 5 days/week

SUMMARY:
This study will evaluate whether a reduction in the radiation dose and field size will maintain a high rate of local control while minimizing the risk of acute and late toxicity.

Hypothesis- The radiation dose and treatment volume can be safely reduced from 30 Gy to 20 Gy while maintaining high rates of local control in patients who had a negative PET scan following rituximab-containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of diffuse large B-cell lymphoma, or any of its variants as defined in the WHO classification
* Completion of at least 4 cycles of a rituximab-containing, anthracycline-based combination chemotherapy
* Negative post-chemotherapy (or interim) PET scan
* Absolute neutrophil count greater than 1500 and platelet count greater than 40,000
* Negative pregnancy test in women of child-bearing potential

For patients with HIV/AIDS, the following must be true:

* The patient is compliant on combination anti-retroviral therapy (CART)
* The patient has CD4 count ≥ 200 at time of diagnosis

Exclusion Criteria:

* Any contraindications to irradiation
* Primary CNS lymphoma
* HIV/AIDS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-09-20 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kelsey, MD, Principal Investigator — Duke University Medical Center, Radiation Oncology
Locations (3):
- United States (3):
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 63
Completed | 62
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 63
Age, Continuous [Median (Full Range); unit: years] | 58 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 52
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Control
Description: This trial will accrue 62 patients over a time period of approximately 5-6 years. The primary objective is to determine whether the number of participants with local control at 5 years, estimated from the Kaplan-Meier curve of time-to-local failure, is as high as that observed in historical controls, i.e., 0.90.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
Participants | 61

2. Secondary Outcome: Percentage of Participants With Progression-free Survival at 5 Years
Description: Progression-free survival (PFS) will be defined as the time from on-study to disease progression or death due to any cause, whichever comes first.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
percentage of participants | 83 [67 to 93]

3. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival will be defined as the number of participants who are alive
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
percentage of participants | 90 [73 to 98]

4. Secondary Outcome: Number of Participants With Local, Distant, or Local+Distant Failure
Description: To examine the patterns of failure, we will tabulate the various ways that patients failed up until the time of the analysis. For example, these ways will include local only, local + distant, and distant only.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
Participants
  Local failure | 1
  Distant failure | 6
  Local+distant failure | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/63
Serious Adverse Events (participants affected / at risk) | 4/63
Other Adverse Events (participants affected / at risk) | 16/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=63)
Papillary thyroid cancer (Endocrine disorders) | 1
Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 2
Papillary carcinoma of the kidney (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=63)
Ear fullness (Ear and labyrinth disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 4
Odynophagia (Gastrointestinal disorders) | 2
Dysgeusia (General disorders) | 1
Gastroesophageal reflux (Gastrointestinal disorders) | 1
Oral mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Idiopathic cardiomyopathy (Cardiac disorders) | 1
Depressed ejection fraction (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT01186978/Prot_SAP_000.pdf